CLINICAL TRIAL: NCT01477697
Title: Effects of Omega-3 Fatty Acid Supplementation on Inflammatory Response in Multisystem Trauma Patients
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Terminated due to slow enrollment and interim analysis showing no difference between treatment arms.
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Krishna Athota, Assistant Clinical Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Athota-2010-01
Record Dates: First submitted 2011-11-18; First posted 2011-11-22 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Multiple Trauma
Keywords: Trauma
MeSH Terms: conditions — Multiple Trauma; Wounds and Injuries | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omega-3 (Active Comparator): 50 mg/kg per day of omega-3 fatty acids (DHA Omega-3, Martek Biosciences, Columbia, MD)
  Interventions: Dietary Supplement: Omega-3
- Placebo (Placebo Comparator): 50 mg/kg per day of vehicle
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Omega-3 — 50 mg/kg per day of omega-3 fatty acids
  Arms: Omega-3
Dietary Supplement: Placebo — 50 mg/kg per day of placebo equivalent
  Arms: Placebo

SUMMARY:
This study will evaluate the effects of omega-3 fatty acid supplementation on inflammation in trauma patients. The main hypothesis is that such supplementation will reduce the presence of biomarkers of systemic inflammation, as compared to placebo

DETAILED DESCRIPTION:
This prospective, randomized study will evaluate the effects of omega-3 fatty acid supplementation on inflammatory response in multi-injured trauma patients. Its primary objective is to compare the intensity of inflammation between an active omega-3 group and a placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Multi-system blunt trauma patients
* Ages 18 through 65 years, inclusive
* Admission to ICU
* Nasogastric or nasoenteric feeding tube in place
* Intention of primary medical team to feed the patient enterally

Exclusion Criteria:

* Expected mortality within 48 hours
* Intracranial hemorrhage
* Pregnant or breast feeding
* Patient, surrogate, or physician not committed to full support
* Refractory shock
* Unable to obtain enteral access
* Presence of partial or complete mechanical bowel obstruction, or ischemia, or infarction
* Current total parenteral nutrition (TPN) use, or intent to use TPN within 7 days
* Current gastrointestinal bleeding
* Requirement for vasopressors

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-06; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Inflammatory markers | Up to 28 days
  Plasma levels of pro-inflammatory cytokines IL-6 and IL-8, as well as C-reactive protein

SECONDARY OUTCOMES:
Infectious complications | Up to 28 days
  Incidence of infectious disease complications using established diagnostic criteria
Intensive Care Unit length of stay | Up to 28 days
  A count of the number of days during which patients are resident in the Surgical Intensive Care Unit

CONTACTS AND LOCATIONS:
Overall Officials: Krishna Athota, MD, Principal Investigator — University of Cincinnati; Richard Branson, MSc, Study Director — University of Cincinnati
Locations (1):
- University Hospital, Cincinnati, Ohio, United States